CLINICAL TRIAL: NCT00250237
Title: Randomised Double-blind Placebo-controlled Study of Post-operative Haloperidol Versus Placebo for Prevention of Post-operative Delirium After Acute Hip Surgery
Brief Title: Post-operative Haloperidol Versus Placebo for Prevention of Post-operative Delirium After Acute Hip Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bronovo Hospital (Other)
Responsible Party: Department of Surgery, Bronovo Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 05-56
Record Dates: First submitted 2005-11-07; First posted 2005-11-08 (Estimated); Last update posted 2009-08-07 (Estimated); Status verified 2009-08

CONDITIONS: Post-Operative Delirium; Hip Fracture
Keywords: Post-operative delirium; hip fracture
MeSH Terms: conditions — Emergence Delirium; Hip Fractures | interventions — Haloperidol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Patients receiving blinded medication (Haloperidol or Placebo)
  Interventions: Drug: Haloperidol
- B (Placebo Comparator): Patients receiving blinded medication (Haloperidol or Placebo)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Haloperidol — Haloperidol 1mg twice daily during 72hours
  Arms: A
Drug: placebo — Placebo 1mg twice daily during 72hours
  Arms: B

SUMMARY:
In this study the investigators want to determine if treatment with haloperidol direct post-operatively after acute hip surgery in high risk patients protects against developing a post-operative delirium.

DETAILED DESCRIPTION:
A post-operative delirium is a serious and frequent (35-65%) complication with high morbidity and mortality in high risk patients. In this study we investigate whether we can prevent a delirium from occuring after surgery in patients with a hip fracture of 75 years of age and older. It's a randomised double-blind single centre placebo-controlled study of haloperidol versus placebo.

ELIGIBILITY:
Inclusion Criteria:

* Hip fracture
* 75 years and older

Exclusion Criteria:

* Contra-indications for the use of haloperidol
* Pre-operative delirium
* Pre-operative use of haloperidol

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 220 (Actual)
Dates: Start 2005-11; Primary Completion 2008-11 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Incidence of post-operative delirium | 72 hours post surgery

SECONDARY OUTCOMES:
Length of stay | days
Complications | during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Boke Linso Sjirk Borger van der Burg, MD, Principal Investigator — Bronovo Hospital
Locations (1):
- Bronovo Hospital, The Hague, South Holland, Netherlands